CLINICAL TRIAL: NCT03037970
Title: A Prospective Randomized Controlled Blinded Study to Evaluate the Safety and Efficacy of rhPDGF-BB Saturated Collagen Wound Dressings on Diabetic Foot Ulcers
Brief Title: Evaluation of ABSOLVE in Diabetic Foot Ulcers
Acronym: ABSOLVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lynch Biologics LLC (Industry)
Collaborators: Medelis Inc. (Industry); Centro Medico Militar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lynch 02-01
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Becaplermin

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, two-arm, clinical study
Who Masked: Participant, Investigator
Masking Description: One component of the study drug will be blinded as the study employs a placebo-controlled arm. More specifically, vials containing rhPDGF or saline will be the same Type I, sodium borosilicate vials with rubber stopper, and plastic cap. Each vial will contain 3 ml of clear liquid. The vials will have blinded labels. Type I collagen wound dressings, on the other hand, will all be the same and are not part of the blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABSOLVE (Experimental): Type I collagen sheet soaked in a solution containing rhPDGF-BB.
  Interventions: Drug: RhPDGF-BB
- Placebo (Placebo Comparator): Collagen sheet soaked with saline solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RhPDGF-BB — One 2x4x.3cm of collagen wound matrix is saturated with 2.0 ml of the rhPDGF-BB solution.
  Other Names: ABSOLVE
  Arms: ABSOLVE
Other: Placebo — Collagen Wound Dressing wetted with buffer.
  Arms: Placebo

SUMMARY:
ABSOLVE Biologic Wound Matrix is a combination of recombinant human platelet-derived growth factor BB homodimer (rhPDGF-BB) and a bovine type I collagen wound dressing matrix. ABSOLVE is under development for the treatment of chronic and acute wounds. This study investigates the safety and efficacy of ABSOLVE in chronic diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
Patients with diabetes are at risk for developing serious health problems that may affect the feet, eyes, kidneys, skin and heart. Foot ulcerations are of great significance to the lives of millions of diabetic patients, representing one of the most common and serious complications in these patients. Up to 25% of diabetics will develop a diabetic foot ulcer (DFU) at some point in their lifetime. The prevalence of DFUs among diabetics is 4% to 10%. More than half of all foot ulcers will become infected requiring hospitalization and 1 in 5 will require amputation. Foot ulcers account for 85,000 non-trauma related lower limb amputations annually in the USA. Every 20 seconds, somewhere in the world, a limb is lost as a consequence of diabetes. Moreover, 85% of leg amputations are preceded by DFUs and more than 60% of non-traumatic lower extremity amputations (LEA) performed in the United States each year occurs secondary to complications of diabetes mellitus. After a major amputation, 50% of patients will have another limb amputated within two years. Mortality rates subsequent to amputation are alarmingly high - up to 40% at 1 year and 80% at 5 years. Patients with a history of a DFU have a 40% greater mortality rate compared to patients with diabetes alone. Improved treatments for DFUs are clearly a matter of great significance.

In this study, the investigation will be focused on the safety and efficacy of ABSOLVE in treating diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adults 30 to 75 years of age
* A diagnosis of Type 1 or 2 diabetes with HbAlc between 6 and 12%, an adequate blood supply defined as TcpO2 > 30 mmHg or an ankle brachial index (ABI) ≥ 0.7 on the foot with the target ulcer
* A DFU 2 cm2-14 cm2 that extends into the subcutaneous tissues or beyond (≤Wagner Grade 2)
* A DFU of at least 6 weeks duration and under care of the study investigator for at least 2 weeks following standard wound debridement with less than 30% healing
* Body Mass Index (BMI) of 18.5 to 40 kg/m2
* Co-morbidities are under control and non-life threatening as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory tests
* A negative pregnancy test at Screening
* Both males and WCBP agree to use acceptable contraceptive methods while on study
* Able to comprehend and sign an ICF.

Exclusion Criteria:

* Evidence of clinically significant findings on screening evaluations (clinical, laboratory, and ECG) which, in the opinion of the Investigator would pose a safety risk or interfere with interpretation of safety data
* Current or recent history of significant bacterial, fungal, viral, or mycobacterial infection
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
* History of myocardial infarction, congestive heart failure, or stroke
* History of psychotic disorder
* History of alcoholism or drug addiction
* Positive drug screen at Screening
* Current treatment or treatment within 30 days prior to first dose of study products with another investigational drug or current enrollment in another clinical trial
* Known history of HIV, hepatitis B, or hepatitis C
* Known hypersensitivity to any of the product's components
* Subjects who are unable or unlikely to comply with the protocol
* Pregnant or lactating.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-30 (Estimated); Primary Completion 2017-08-15 (Estimated); Study Completion 2017-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Week 0 - 24
  Determine safety and tolerability of ABSOLVE on patients having a poorly healing diabetic foot ulcer.
Successful wound healing for at least two consecutive measurements. (Efficacy) | Week 12
  Successfully healed wound must remain closed for at least two consecutive measurements, one of which will be at the 12-week examination.

SECONDARY OUTCOMES:
Wound Size | Week 0 - 24
  The percent change in wound size (closure) over time.
Wound Closure | Week 0 - 24
  Percent incidence of complete wound closure over time.
Complication rate | Week 0 - 24
  Reduction in complications.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Gonzalez, MD, Principal Investigator — Centro Medico Militar, Guatemala
Locations (1):
- Centro Medico Militar, Guatemala City, Guatemala

IPD SHARING:
Plan to Share IPD: Undecided